CLINICAL TRIAL: NCT03779906
Title: A Prospective, Multicenter Observational Study to Evaluate Thyroid Function of Pediatric Subjects From Birth to 3 Years Exposed to ISOVUE® (Iopamidol Injection)
Brief Title: Thyroid Function of Pediatric Subjects Following Isovue® Administration
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Formal release from PMR
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IOP-120
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hypothyroidism
Keywords: hypothyroidism; ISOVUE; Iodinated Contrast Agent
MeSH Terms: conditions — Hypothyroidism | interventions — Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ISOVUE (Experimental): Isovue will be given to all subjects per the standard of clinical care.The specific iodine concentration and volume of ISOVUE used during the radiologic procedure will depend on the type of procedure and the standards in place at the site where the procedure is performed.
  Interventions: Drug: Isovue

INTERVENTIONS:
Drug: Isovue — Isovue will be given to all subjects per the standard of clinical care.
  Other Names: IOPAMIDOL injection

SUMMARY:
This is a Phase IV prospective, multicenter, observational study to estimate the proportion of subjects 0 to 3 years of age who develop abnormal thyroid function after exposure to intravascular administration of ISOVUE for the required radiologic procedure as part of their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female from 0 to 3 years of age;
* Is scheduled to undergo a radiologic examination that requires intravascular administration of ISOVUE as part of his/her standard of care;
* Has normal baseline thyroid function tests (TSH, total T3, total T4, and fT4) performed at a local laboratory with blood sample obtained within one week prior to ISOVUE administration;
* Written informed consent is obtained from the subject's parent(s) or legally acceptable representative(s) (according to local regulations) who are willing to comply with the protocol requirements.

Exclusion Criteria:

* Has any known allergy to one or more of the ingredients of ISOVUE;
* Has been diagnosed with congenital hypothyroidism;
* Has undergone radiation treatments to the head or neck;
* Is currently on thyroid replacement therapy;
* Is on therapy with dopamine or any treatment which may affect the thyroid function testing results;
* Has been exposed to any topical iodinated product within 30 days prior to enrollment in the present study;
* Has been exposed to an iodinated contrast agent within 1 year prior to enrollment in the present study, including any administration of iodinated contrast agents during placement of a central line;
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Luigia Storto, MD, Study Director — Bracco Corporate
Locations (4):
- United States (4):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On 03 March 2022, Food and Drug Administration (FDA) released Bracco from the Post-Marketing Requirement (PMR) commitment as the risk of thyroid dysfunction was adequately addressed by FDA's review of findings reported in currently available publications. Therefore, the study was terminated on 25 March 2022 with only 17 subjects enrolled and dosed.
Pre-assignment Details: Pediatric subjects (0-3 years of age) scheduled to undergo a routine radiologic procedure with intravascular administration of ISOVUE who had normal TFTs (serum TSH, T3, T4 & fT4) at baseline were to be enrolled. TFTs were to be reassessed at 1 month and 2 months post-ISOVUE injection. If TSH values were abnormal at 1- or 2-months, follow-up (via pre-defined questionnaire) was required at 6 and 12 months to monitor subject's progress (if any). Efficacy of ISOVUE was not assessed.
Groups:
- ISOVUE: Intravascular administration of ISOVUE as part of the subject's standard of care examination.
Period: Overall Study
Arm/Group | ISOVUE
Started | 17
Completed | 9
Not Completed | 8
Not completed — Lost to Follow-up | 7
Not completed — COVID pandemic | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled and dosed in the study who provided demographic information.
Arm/Group | ISOVUE
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  Between 0 to 3 years | 17
  Between 4 to 17 years | 0
  Between 18 and 65 years | 0
  Above 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  Black | 2
  Latino | 1
  More than one race | 1
Region of Enrollment [Number; unit: participants]
  United States | 17
Number of Subjects with TFTs at Baseline [Count of Participants; unit: Participants]
  Normal | 17
  Abnormal | 0

OUTCOME MEASURES:

1. Primary Outcome: Abnormal Thyroid Function
Description: The primary outcome of this study was to evaluate the proportion of subjects, 0 to 3 years of age, with abnormal TSH values post-baseline following administration of ISOVUE.
Time Frame: Day 1 (day dosed with intravascular administration of ISOVUE as part of their standard of care examination) to 1-month follow-up or 2-month follow-up
Population: Number of subjects evaluated for TFTs at baseline and post-baseline following intravascular administration of ISOVUE.
Measure: Count of Participants; unit: Participants
Groups:
- ISOVUE: Intravascular administration of ISOVUE as part of a subject's standard of care examination.
Arm/Group | ISOVUE
Number analyzed (Participants) | 17
Participants
  Number of Patients with Abnormal TSH only at 1-month follow-up | 0
  Number of Patients with Abnormal TSH only at 2-month follow-up | 0
  Number of Patients with Abnormal TSH at 1 and 2 months' follow-up | 0
  Number of Patients with Normal TSH at All Follow-up Timepoints | 17

2. Secondary Outcome: Hypothyroidism
Description: To evaluate the proportion of subjects, 0 to 3 years of age, with hypothyroidism regardless of the need for thyroid hormone therapy after administration of ISOVUE.
Time Frame: as for outcome 1
Population: Number of subjects evaluated for TFTs at baseline and post-baseline following intravascular administration of ISOVUE.
Measure: Count of Participants; unit: Participants
Arm/Group | ISOVUE
Number analyzed (Participants) | 17
Participants
  Number of subjects with hypothyroidism at 1-month follow-up | 0
  Number of subjects with hypothyroidism at 2-month follow-up | 0
  Number of subjects with normal thyroid values through 2-month follow-up | 17

3. Secondary Outcome: Thyroid Hormone Replacement Therapy
Description: The proportion of subjects initiated on thyroid hormone replacement therapy.
Time Frame: Day 1 (day dosed with intravascular administration of ISOVUE as part of their standard of care examination) to 1-month follow-up or 2-month follow-up to 6- to 12 months follow-up (if applicable)
Population: Number of subjects evaluated for TFTs at baseline and post-baseline following intravascular administration of ISOVUE.
Measure: Count of Participants; unit: Participants
Arm/Group | ISOVUE
Number analyzed (Participants) | 17
Participants
  Number of subjects who started hormone therapy by 1-month follow-up | 0
  Number of subjects who started hormone therapy by 2-month follow-up | 0
  Number of subjects who did not start hormone therapy through 2-month follow-up | 17
  Number of subjects who started hormone therapy by 6- or 12-month follow-up | NA — Subjects were not further evaluated at 6 and 12 months if there were no abnormal TSH values at 1 and/or 2 months follow-up.

ADVERSE EVENTS:
Time Frame: As this was an Observational Study, untoward medical occurrences (i.e., adverse events) were monitored through completion of the exam with administration of ISOVUE, up to 1 week for subjects dosed as part of their routine standard of care.
Description: Subjects were monitored for any untoward medical occurrences from the time of signed Informed Consent through the timeframe associated with the investigational medicinal product administration. All untoward medical occurrences were recorded in the Adverse Event section of the CRF.
Arm/Group | ISOVUE
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISOVUE (N=17)
Pyrexia (General disorders) | 1 (1) — fever, occurred 7 days postdose, no reasonable possibility of relationship to administration of investigational product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT03779906/Prot_000.pdf